CLINICAL TRIAL: NCT06675994
Title: Evaluation of PCSK9 Enzyme in Non-Cholesterol Biological Pathways: In Vitro Demonstration of Direct Platelet-Related Effects of PCSK9 Enzyme
Brief Title: In Vitro Demonstration of Direct Platelet-Related Effects of PCSK9 Enzyme
Status: Not yet recruiting | Type: Observational
Sponsor: LifeBridge Health (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Paul A. Gurbel, Director of Cardiovascular Research, LifeBridge Health
Other Study IDs: 2253810
Record Dates: First submitted 2024-11-01; First posted 2024-11-06 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Healthy; Hypercholesterolemia; Hypertension; Overweight; Prediabetes; Diabetes; Family History of Coronary Artery Disease; Family History of Peripheral Artery Disease; Family History of Cerebrovascular Disease
MeSH Terms: conditions — Hypercholesterolemia; Hypertension; Overweight; Prediabetic State; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Healthy: Participants (approximately 40) 18-50 years old male and female without any major medical conditions or taking any agents or food supplements that may influence platelet function as determined by the study principal investigator.
  Interventions: Drug: PCSK9 Antibody, PCSK9 Enzyme
- Cardiovascular Risk Factor: Participants (approximately 40) 18-50 years old male and female with at least three of the following risk factors: history of hypercholesterolemia, hypertension, overweight, current smoker, prediabetes or diabetes who are only on metformin and insulin, and a family history of coronary artery, peripheral artery, or cerebrovascular disease.
  Interventions: Drug: PCSK9 Antibody, PCSK9 Enzyme

INTERVENTIONS:
Drug: PCSK9 Antibody, PCSK9 Enzyme — In-vitro demonstration of the direct effect if the PCSK9 enzyme on platelets. The study will use commercially available recombinant PCSK9 enzyme to promote platelet activity and the PCSK9 antibody to inhibit activity. In each patient, platelet function testing will occur in the absence of PCSK9 enzyme, after the addition of PCSK9 enzyme, and after the addition of both PCSK9 enzyme and antibody reagent to the blood sample prior to testing.

SUMMARY:
Proprotein convertase subtilisin/kexin type 9 (PCSK9) has evolved as a pivotal enzyme in lipid metabolism and therapeutic target for hypercholesterolemia and atherosclerotic cardiovascular disease (CVD). Furthermore, research from in-vitro and in-vivo animal models suggest that the inhibition of PCSK9 expression may suppress platelet activation, and systemic inflammation thereby reducing thrombotic risk. Taken together, these data support the lower rates of myocardial infarction, stroke, and coronary revascularization in subjects with increased CVD risk in clinical trials with alirocumab (Praluent) and evolocumab (Repatha) as compared to placebo. The main aim of this single center, exploratory in-vitro evaluation is to investigate the direct role of PCSK9 on platelet activation and aggregation using blood collected from a diverse population of antiplatelet naïve healthy volunteers (n=40) and subjects with CVD risk factors (n=40) between the 18-50 years of age. All procedures including consenting, collection of clinical data, and lab processing will occur at the Sinai Center for Thrombosis Research. The results of this study will provide a better understanding of cardioprotective effects of PCSK9 inhibition beyond lipid lowering.

DETAILED DESCRIPTION:
The pivotal role of platelets during arterial ischemic events, such as myocardial infarction (MI), stroke, and cardiovascular (CV) death, and the significant role of potent antiplatelet therapy in reducing these events have been well defined. An independent association between plasma PCSK9 levels, elevated platelet reactivity, and ischemic outcomes in patients with acute coronary syndromes (ACS) has been demonstrated. The association of plasma PCSK9 levels with coronary artery disease (CAD) risk, independent of low-density lipoprotein cholesterol (LDL-C) levels, has been suggested. Based on a meta-analysis of trials of medium-high risk cardiovascular disease (CVD) patients, the investigators have demonstrated a significant mortality and MI reduction with PCSK9 antibodies and suggested a relevant ant ischemic/antiplatelet role of PCSK9 antibodies. These observations support the hypothesis that the anti-ischemic effects of PCSK9 inhibitor therapy are related to its pleiotropic effects on platelets.

In vitro, animal, and human studies have suggested the direct effects of PCSK9 and PCSK9 inhibitors on platelets. PCSK9 indirectly activates platelets through elevated LDL-C and oxLDL levels. oxLDL can activate platelets by binding to the scavenger receptors CD36 and LOX-1. In addition, a direct relationship between PCSK9 and platelet activation through the scavenger receptors CD36 and Lectin-like oxidized LDL receptor (LOX)-1 has been suggested. Incubation of human recombinant PCSK9 protein with platelet-rich plasma collected from healthy subjects significantly enhanced activated GPIIb/IIIa receptor expression and platelet aggregation induced by suboptimal concentrations of epinephrine. In in vitro experiments, human recombinant PCSK9 exposure enhanced LOX-1 expression in human vascular endothelial cells and smooth muscle cells. Similarly, LOX-1 KO mice showed lower PCSK9 levels and PCSK9-KO mice showed much lower LOX-1 levels, indicating a reciprocal relationship between PCSK9 and LOX-1. A similar reciprocal relationship between PCSK9 levels and LOX-1 and CD36 expression has not been demonstrated in human platelets.

In vitro immunoblotting experiments demonstrated the presence of PCSK9 in platelets obtained from patients with CAD, and flow cytometry experiments demonstrated that collagen-related peptide (CP) significantly enhanced the surface expression of PCSK9 on platelets. Furthermore, PCSK9 antibodies significantly inhibited ADP- and CP-induced platelet aggregation and platelet-dependent thrombus formation on the immobilized collagen surface under high shear rate (1000s-1). Binding of PCSK9 to CD36 triggers platelet activation through activation of nicotinamide adenine dinucleotide phosphate oxidase (Nox)2, release of reactive oxygen species (ROS), and subsequent activation of GPIIb/IIIa receptor and p-selectin release. In addition, Nox2 induces the generation of 8-Iso-prostaglandin F2α and thromboxane (Tx) A2 through the activation f cytosolic phospholipase A2 and finally results in the activation of the GP-IIb/IIIa receptor and p-selectin release. The relationship between plasma PCSK9, urinary 11-dehydro-TxB2, and CV events in patients with atrial fibrillation has been demonstrated. Furthermore, washed platelets resuspended in plasma from patients with familial hypercholesterolemia after PCSK9 inhibitor treatment induced lower platelet aggregation and soluble Nox2-derived peptide (sNox2-dp) release than those obtained using plasma before PCSK9 inhibitor treatment in an in vitro study. This reduction was reversed by the addition of oxLDL. Furthermore, oxLDL-induced platelet aggregation was reduced by inhibiting CD36, LOX-1, and Nox2. In the same study, 6-month treatment with PCSK9 inhibitors was shown to reduce serum LDL-C, oxLDL, serum TxB2, sNox2-dp, and PCSK9 levels.

These preliminary observations suggest that:

* CV benefits associated with PCSK9 inhibitor therapy may be in part related to its pleiotropic effects on platelets.
* In vitro, animal, and clinical studies suggested direct effects of PCSK9 on platelets.
* PCSK9 influence platelet function through CD36/LOX-1 receptor mediated Nox2 activity.

However, the potential direct platelet effects of PCSK9 on platelets have not been demonstrated in a comprehensive study involving a diverse population of healthy volunteers and subjects with cardiovascular risk factors. Inclusion of at least 3 CV risk factors will increase the chance of finding subjects with an elevated platelet reactivity phenotype and demonstration of enhanced platelet-related effect of PCSK9. The presence of these risk factors has been traditionally attributed to increased prevalence of CVD and associated risk.

In contemporary CV clinical trials, a very low percentage (<10%) of African Americans are represented despite a more pronounced CVD risk. Furthermore, it has been demonstrated that PCSK9 levels are significantly higher in African Americans vs Caucasians (104 ± 29 vs 95 ± 30 ng/mL, respectively; P = 0.020). At Sinai Hospital of Baltimore, the investigators have reported higher rates of post-PCI ischemic events and greater mortality in African Americans than in Whites. Rare loss-of-function (LoF) mutations of PCSK9 have been associated with low levels of LDL-C (28% lower in Blacks and 15% in Whites) and with an even more impressive reduction in the risk of coronary artery disease (CAD) (88% and 47%, respectively). PCSK9 LoF variants were associated with 35 mg/dL and 13 mg/dL lower LDL-C levels in African Americans and Caucasians, respectively, and a 49% and 18% lower risk for coronary heart disease in African Americans and Caucasians, respectively. In a study of 10,196 US African American adults, PCSK9 LoF variants were associated with lower concentrations of lipoprotein (Lpa) and OxPL-apoB. These data indicate a direct relationship between PCSK9 and the risk of CAD, and the importance of lowering PCSK9 levels in reducing CAD risk among African Americans.

The knowledge gained by our exploratory mechanistic study will help us to understand the direct effects of PCSK9 and PCSK9 inhibitor on platelets and facilitate the clinical application of PCSK9 inhibitors in a broad range of patients with cardiovascular risk.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects (n=40): 18-50 years old male and female subjects without any conditions or taking any agents or food supplements that may influence platelet function as determined by the study principal investigator.
* Subjects with CV risk factors (n=40): 18-50 years old male and female subjects with at least three of the following CV risk factors:

History of hypercholesterolemia, hypertension, overweight, current smoker, prediabetes or diabetes who are only on metformin and insulin, and family history of coronary artery, peripheral artery, or cerebrovascular disease.

Overweight is defined as subjects with BMI ≥25 kg/m2 (https://www.heart.org/en/healthy-living/healthy-eating/losing-weight/bmi-in-adults).

Diabetes is defined as haemoglobin (Hb)A1c ≥6.5%, prediabetes =5.7%-6.4%) (https://diabetes.org/about-diabetes/diagnosis)

Exclusion Criteria:

* Subjects with Diabetes mellitus, who are on GLP-1 agonists or SGLT2 inhibitors.
* Subjects on high dose statin therapy or PCSK9 therapy.
* Prior coronary of cerebrovascular event requiring intervention.
* Use of any antiplatelet or anticoagulant therapy within 14 days of enrollment.
* Subjects with a history of chronic kidney disease, liver disease, pancreatitis, HIV, hepatitis, and active cancer, active infection, or any other medical condition or concomitant medications as determined by the investigator that may affect study results.
* Pregnant

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This trial has been designed to ensure enrollment of healthy volunteers and subjects with CV risk to allow for comparisons across disease states in order to fulfill study objectives. Compared to healthy volunteers, subjects with CV risk factors are highly prothrombotic and exhibit a high platelet reactivity phenotype. Coexistence of at least three risk factors indicate a high risk for future CV events. African Americans and women are inherently at elevated risk for CVD, associated ischemic events, and exhibit higher serum PCSK9 levels. Therefore, equal inclusion of race and genders should provide robust variability in PCSK9 levels for evaluation of platelet related effects of PCSK9.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Difference in ADP-induced platelet aggregation (%) with and without PCSK9 enzyme | Throughout study completion, an average of about 1 year
  Difference in ADP-induced platelet aggregation (%) with and without addition of PCSK9 enzyme in blood collected from healthy volunteers and subjects with cardiovascular risk factors.
Difference in collagen related peptide -induced platelet aggregation (%) with and without PCSK9 enzyme | Throughout study completion, an average of about 1 year
  Difference in collagen related peptide-induced platelet aggregation (%) with and without PCSK9 enzyme in blood collected from healthy volunteers and subjects with cardiovascular risk factors.

SECONDARY OUTCOMES:
Difference in ADP-induced platelet aggregation (%) with PCSK9 enzyme alone and with addition of PCSK9 antibody | Throughout study completion, an average of about 1 year
  Difference in ADP-induced platelet aggregation (%) with PCSK9 enzyme alone and after addition of PCSK9 antibody in blood collected from healthy volunteers and subjects with cardiovascular risk factors
Difference in collagen related peptide-induced platelet aggregation (%) with PCSK9 enzyme alone and with addition of PCSK9 antibody | Throughout study completion, an average of about 1 year
  Difference in collagen related peptide-induced platelet aggregation (%) with PCSK9 enzyme alone and with addition of PCSK9 antibody in blood collected from healthy volunteers and subjects with cardiovascular risk factors.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Gurbel, MD, FACC, Principal Investigator — LifeBridge Health

IPD SHARING:
Plan to Share IPD: Undecided
This is an exploratory in-vitro study not involving clinical outcome endpoints and may not necessitate sharing individual data. A decision will be made after the study is underway.

REFERENCES:
- [Background] Gurbel PA, Tantry US. Combination antithrombotic therapies. Circulation. 2010 Feb 2;121(4):569-83. doi: 10.1161/CIRCULATIONAHA.109.853085. No abstract available. PMID 20124137
- [Background] Gurbel PA, Fox KAA, Tantry US, Ten Cate H, Weitz JI. Combination Antiplatelet and Oral Anticoagulant Therapy in Patients With Coronary and Peripheral Artery Disease. Circulation. 2019 Apr 30;139(18):2170-2185. doi: 10.1161/CIRCULATIONAHA.118.033580. PMID 31034291
- [Background] Navarese EP, Kolodziejczak M, Winter MP, Alimohammadi A, Lang IM, Buffon A, Lip GY, Siller-Matula JM. Association of PCSK9 with platelet reactivity in patients with acute coronary syndrome treated with prasugrel or ticagrelor: The PCSK9-REACT study. Int J Cardiol. 2017 Jan 15;227:644-649. doi: 10.1016/j.ijcard.2016.10.084. Epub 2016 Oct 29. PMID 27810295
- [Background] Leander K, Malarstig A, Van't Hooft FM, Hyde C, Hellenius ML, Troutt JS, Konrad RJ, Ohrvik J, Hamsten A, de Faire U. Circulating Proprotein Convertase Subtilisin/Kexin Type 9 (PCSK9) Predicts Future Risk of Cardiovascular Events Independently of Established Risk Factors. Circulation. 2016 Mar 29;133(13):1230-9. doi: 10.1161/CIRCULATIONAHA.115.018531. Epub 2016 Feb 19. PMID 26896437
- [Background] Ding Z, Liu S, Wang X, Deng X, Fan Y, Shahanawaz J, Shmookler Reis RJ, Varughese KI, Sawamura T, Mehta JL. Cross-talk between LOX-1 and PCSK9 in vascular tissues. Cardiovasc Res. 2015 Sep 1;107(4):556-67. doi: 10.1093/cvr/cvv178. Epub 2015 Jun 19. PMID 26092101
- [Background] Camera M, Rossetti L, Barbieri SS, Zanotti I, Canciani B, Trabattoni D, Ruscica M, Tremoli E, Ferri N. PCSK9 as a Positive Modulator of Platelet Activation. J Am Coll Cardiol. 2018 Feb 27;71(8):952-954. doi: 10.1016/j.jacc.2017.11.069. No abstract available. PMID 29471945
- [Background] Petersen-Uribe A, Kremser M, Rohlfing AK, Castor T, Kolb K, Dicenta V, Emschermann F, Li B, Borst O, Rath D, Muller KAL, Gawaz MP. Platelet-Derived PCSK9 Is Associated with LDL Metabolism and Modulates Atherothrombotic Mechanisms in Coronary Artery Disease. Int J Mol Sci. 2021 Oct 16;22(20):11179. doi: 10.3390/ijms222011179. PMID 34681838
- [Background] 15. Pastori D, Nocella C, Farcomeni A, et al. ATHERO-AF Study Group. Relationship of PCSK9 and Urinary Thromboxane Excretion to Cardiovascular Events in Patients With Atrial Fibrillation. J Am Coll Cardiol. 2017 Sep 19;70(12):1455-1462. doi: 10.1016/j.jacc.2017.07.743. PMID: 28911508. Cammisotto V, Pastori D, Nocella C, et al. PCSK9 Regulates Nox2-Mediated Platelet Activation via CD36 Receptor in Patients with Atrial Fibrillation. Antioxidants (Basel). 2020;9:296.
- [Background] Cammisotto V, Pastori D, Nocella C, Bartimoccia S, Castellani V, Marchese C, Scavalli AS, Ettorre E, Viceconte N, Violi F, Pignatelli P, Carnevale R. PCSK9 Regulates Nox2-Mediated Platelet Activation via CD36 Receptor in Patients with Atrial Fibrillation. Antioxidants (Basel). 2020 Apr 2;9(4):296. doi: 10.3390/antiox9040296. PMID 32252393
- [Background] Tsao CW, Aday AW, Almarzooq ZI, Alonso A, Beaton AZ, Bittencourt MS, Boehme AK, Buxton AE, Carson AP, Commodore-Mensah Y, Elkind MSV, Evenson KR, Eze-Nliam C, Ferguson JF, Generoso G, Ho JE, Kalani R, Khan SS, Kissela BM, Knutson KL, Levine DA, Lewis TT, Liu J, Loop MS, Ma J, Mussolino ME, Navaneethan SD, Perak AM, Poudel R, Rezk-Hanna M, Roth GA, Schroeder EB, Shah SH, Thacker EL, VanWagner LB, Virani SS, Voecks JH, Wang NY, Yaffe K, Martin SS. Heart Disease and Stroke Statistics-2022 Update: A Report From the American Heart Association. Circulation. 2022 Feb 22;145(8):e153-e639. doi: 10.1161/CIR.0000000000001052. Epub 2022 Jan 26. PMID 35078371
- [Background] Gerstein HC, Branch K, Heenan L, Del Prato S, Khurmi NS, Lam CSP, Pratley R, Rosenstock J, Sattar N. Design and baseline characteristics of the AMPLITUDE-O cardiovascular outcomes trial of efpeglenatide, a weekly glucagon-like peptide-1 receptor agonist. Diabetes Obes Metab. 2021 Feb;23(2):318-323. doi: 10.1111/dom.14223. Epub 2020 Oct 22. PMID 33026143
- [Background] Gurbel PA, Bliden KP, Guyer K, Cho PW, Zaman KA, Kreutz RP, Bassi AK, Tantry US. Platelet reactivity in patients and recurrent events post-stenting: results of the PREPARE POST-STENTING Study. J Am Coll Cardiol. 2005 Nov 15;46(10):1820-6. doi: 10.1016/j.jacc.2005.07.041. Epub 2005 Oct 21. PMID 16286165
- [Background] Lev EI, Bliden KP, Jeong YH, Pandya S, Kang K, Franzese C, Tantry US, Gurbel PA. Influence of race and sex on thrombogenicity in a large cohort of coronary artery disease patients. J Am Heart Assoc. 2014 Oct 20;3(5):e001167. doi: 10.1161/JAHA.114.001167. PMID 25332180
- [Background] Cohen JC, Boerwinkle E, Mosley TH Jr, Hobbs HH. Sequence variations in PCSK9, low LDL, and protection against coronary heart disease. N Engl J Med. 2006 Mar 23;354(12):1264-72. doi: 10.1056/NEJMoa054013. PMID 16554528
- [Background] Kent ST, Rosenson RS, Avery CL, Chen YI, Correa A, Cummings SR, Cupples LA, Cushman M, Evans DS, Gudnason V, Harris TB, Howard G, Irvin MR, Judd SE, Jukema JW, Lange L, Levitan EB, Li X, Liu Y, Post WS, Postmus I, Psaty BM, Rotter JI, Safford MM, Sitlani CM, Smith AV, Stewart JD, Trompet S, Sun F, Vasan RS, Woolley JM, Whitsel EA, Wiggins KL, Wilson JG, Muntner P. PCSK9 Loss-of-Function Variants, Low-Density Lipoprotein Cholesterol, and Risk of Coronary Heart Disease and Stroke: Data From 9 Studies of Blacks and Whites. Circ Cardiovasc Genet. 2017 Aug;10(4):e001632. doi: 10.1161/CIRCGENETICS.116.001632. PMID 28768753
- [Background] Mefford MT, Marcovina SM, Bittner V, Cushman M, Brown TM, Farkouh ME, Tsimikas S, Monda KL, Lopez JAG, Muntner P, Rosenson RS. PCSK9 loss-of-function variants and Lp(a) phenotypes among black US adults. J Lipid Res. 2019 Nov;60(11):1946-1952. doi: 10.1194/jlr.P119000173. Epub 2019 Sep 11. PMID 31511398
- [Background] Chaudhary R, Sukhi A, Chaudhary R, Jindal M, Vyas A, Rout A, Bliden K, Tantry U, Gurbel P. Gender differences in thrombogenicity among patients with angina and non-obstructive coronary artery disease. J Thromb Thrombolysis. 2019 Oct;48(3):373-381. doi: 10.1007/s11239-019-01901-1. PMID 31218482